CLINICAL TRIAL: NCT07144267
Title: Milrinone Versus Epinephrine for Right Ventricular Dysfunction After Cardiac Surgery in Adults: A Randomized Double-Blinded Trial
Brief Title: Comparison of Milrinone and Epinephrine on TAPSE
Acronym: Milrinone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Professor of Anesthesia , surgical Intensive care and pain management Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Milrinone on TAPSE
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Anaesthesia; Cardiopulmonary Bypass
Keywords: Cardiopulmonary bypass (CPB) -Tricuspid annular plane systolic excursion (TAPSE)-; Epinephrine - Milrinone
MeSH Terms: interventions — Epinephrine; Milrinone

STUDY DESIGN:
Intervention Model Description: Epinephrine group (group E): the patients receive 0.05-0.1 mcg/kg/min.of epinephrine 5-10 minutes before aortic unclamping.
  Milrinone group (group M): the patients receive initial bolus doses of 50 µg/kg, followed by 0.40 - 0.80 µg/kg/min of milrinone 5-10 minutes before aortic unclamping
Who Masked: Participant, Investigator
Masking Description: anesthesiologist who performed TEE measurements and who was responsible for data collection will be blinded to patient group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Epinephrine group (group E) (Active Comparator): The patients receive 0.05-0.1 mcg/kg/min.of epinephrine 5-10 minutes before aortic unclamping
  Interventions: Drug: Epinephrine
- Milrinone group (group M) (Active Comparator): patients will recieve an initial bolus dose of of 50 µg/kg, followed by 0.40 -0.80 µg/kg/min 5-10 minutes before aortic unclamping
  Interventions: Drug: Milrinone Injection

INTERVENTIONS:
Drug: Epinephrine — Normal saline bolus over 10 min followed by Epinephrine intravenous infusion of 0.05-0.1 mcg/kg/min.of epinephrine 5-10 minutes before aortic unclamping
  Arms: Epinephrine group (group E)
Drug: Milrinone Injection — Milrinone initial bolus doses of 50 µg/kg, followed by 0.40 - 0.80 µg/kg/min of milrinone 5-10 minutes before aortic unclamping
  Arms: Milrinone group (group M)

SUMMARY:
Cardiopulmonary bypass (CPB) is a critical technology in cardiac surgery, allowing for the temporary replacement of the heart and lung functions during intricate surgical procedures. it has significant post-surgical complications, the most important complications of CPB is right ventricle (RV) dysfunction. Diagnosis and management of RV dysfunction is crucial for maintenance of hemodynamic stability and organ function in early post-operation period and prognostic for later phase.

DETAILED DESCRIPTION:
Epinephrine is the most potent adrenergic agonist which has positive inotropic and chronotropic effects and enhanced conduction in the heart (β1), smooth muscle relaxation in the vasculature and bronchial tree (β2), and vasoconstriction (α1). Low doses of this agent (<0.1-0.2 μg/kg/min) mainly activate the β adrenoceptors with inotropic effects. Higher doses result in vasoconstrictor effect which takes the lead. Other effects include bronchial dilation, mydriasis, glycogenolysis, tachyarrhythmia, myocardial ischemia, pulmonary hypertension, hyperglycemia, and lactic acidosis. Epinephrine also reduces splanchnic and hepatic perfusion and increases metabolic workload of the liver. So this hypermetabolism that impairs oxygen exchange, glycolysis, and suppression of insulin cause lactic acidosis.

Milrinone is a phosphodiesterase-III inhibitor. This effect decreases the degradation of cyclic adenosine monophosphate (cAMP), increases the cAMP levels in cells, and then increases activation of protein kinase A. Therefore, its cardiac effects are positive inotropy and improved diastolic relaxation. Milrinone also causes potent vasodilation, with reduction in preload, afterload and pulmonary vascular resistance. Considering its characteristics, milrinone might be a useful agent for cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II & III
* Age between 18 and 70 years
* Both Gender
* Body mass index less than 40 kg/m2
* Ejection fraction of >40%
* Tricuspid annular plane systolic excursion (TAPSE) < 1.7cm

Exclusion Criteria:

* Patient refusal.
* Preoperative RV impairment
* Pulmonary hypertension (estimated pulmonary artery systolic pressure > 50 mmHg)
* Patients with any contraindications to Transesophageal echocardiography (TEE)
* Redo or Re-exploration surgery
* Patients with chronic kidney disease (serum creatinine > 1.5 mg/ dl)
* Patients with chronic liver disease (child pugh B and C)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Tricuspid annular plane systolic excursion (TAPSE) within 5 minutes post-cardiopulmonary Bypass | within 5 mins post-cardiopulmonary bypass
  measured by Transesophageal echocardiography (TEE)

SECONDARY OUTCOMES:
Tricuspid annular plane systolic excursion (TAPSE) | within 30-60 minutes post-cardiopulmonary bypass
  measured by Transesophageal echocardiography (TEE)
Incidence of Right Ventricular Dysfunction after Cardiac Surgery | 24 hours postoperative
  detected by ECHO when Tricuspid annular plane systolic excursion (TAPSE) ≤1.7 cm
Incidence of Arrhythmias | intraoperatively and 24 hours postoperative
  occurrence of any Arrhythmia
Vasoactive-Inotrope Score (VIS) | recorded at 6, 12, 24, and 48 hours postoperative
  Vasoactive-Inotrope Score = Dopamine (µg/kg/min) + Dobutamine (µg/kg/min) +100 x Epinephrine (µg/kg/min) +100 x Norepinephrine (µg/kg/min) + 10 x Milrinone (µg/kg/min) + 10,000 x Vasopressin
Total consumption doses of Vasopressors | 48 hours postoperative
  cumulative dose of any needed Vasopressors (Norepinepherine)